CLINICAL TRIAL: NCT04107766
Title: A Multicenter Observational Registry to Develop Ablation Parameter Guidance for Microwave Liver Ablation of Soft Tissue Lesions
Brief Title: NOLA (NeuWave Observational Liver Ablation) Registry
Status: Terminated | Type: Observational
Why Stopped: Change in Company Strategy
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NEU_2017_04
Record Dates: First submitted 2019-09-05; First posted 2019-09-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer of the Liver; Liver Cancer; Neoplasms, Liver
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Population: Patients with at least one soft-tissue liver lesion ablated with the NEUWAVE Microwave Ablation System or NEUWAVE Microwave Ablation System with Ablation Confirmation.
  Interventions: Device: Microwave Ablation

INTERVENTIONS:
Device: Microwave Ablation — Patients who meet the eligibility criteria will undergo microwave ablation (MWA) with the NEUWAVE Microwave Ablation System with or without Ablation Confirmation of at least one soft-tissue liver lesion, in accordance with the study site's standard-of-care (SOC) practices.

SUMMARY:
This is a multicenter, observational registry that follows patients for a total of 5 years from the date of the first liver ablation procedure with the NEUWAVE Microwave Ablation System.

DETAILED DESCRIPTION:
This is a multicenter, observational registry that follows patients for a total of 5 years from the date of the first liver ablation procedure with the NEUWAVE Microwave Ablation System. The data gathered from participating sites will be available to be analyzed to develop ablation parameter guidance for ablation approaches under varying patient liver tissue conditions and liver lesions.

This is an "umbrella registry," which was included as an optional component in other NEUWAVE studies; hence, data from consenting patients who are or will be enrolled in other NEUWAVE soft tissue liver lesion ablation studies will be included in this registry. All other patients will be enrolled and followed prospectively, enrolled retrospectively with prospective, longitudinal follow up, or enrolled retrospectively with all retrospective follow up.

Enrollment for this study will include up to 1,500 patients throughout the world who underwent or are scheduled to undergo microwave ablation of one or more soft tissue liver lesions using the NEUWAVE Microwave Ablation System or the NEUWAVE Microwave Ablation System with Ablation Confirmation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent or are scheduled to undergo a microwave ablation of one or more liver lesions with the NEUWAVE Microwave Ablation System per the device's Instructions for Use (IFU).
2. Patients with signed informed consent (or waiver approved by IRB/EC) who are willing to comply with the assessment schedule, and willing to have data included in the database.
3. Patients greater than or equal to 22 years old at the time of informed consent (or waiver approved by IRB/EC).

Exclusion Criteria:

1. Patients with a life expectancy of less than 1 year, in the opinion of the treating physician.
2. Use of microwave ablation purely as a transection tool, rather than focused liver lesion ablation.
3. Patient is currently participating, or planning to participate, in another NeuWave/Ethicon-funded clinical trial or registry studying microwave ablation in the liver. Note: roll-over patients from previous NeuWave trials are permitted.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with at least one soft-tissue liver lesion ablated with the NEUWAVE Microwave Ablation System or NEUWAVE Microwave Ablation System with Ablation Confirmation.
Sampling Method: Non-Probability Sample
Enrollment: 1255 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Technical success | Day of ablation (Day 0)
  Technical success, defined as ablation of the target lesion(s) according to the protocol and covered completely, with an adequate margin, as defined by the performing physician (i.e. the ablation zone completely overlaps or encompasses the target lesion(s) plus an ablative margin), as assessed by CT, MRI, PET, US, and/or X-ray, immediately following the procedure.
Technical efficacy | 7 days to 3 months post-ablation
  Technique efficacy, ablation of the target lesion(s) according to the protocol and covered completely, with an adequate margin, as defined by the performing physician (i.e., the ablation zone completely overlaps or encompasses the target lesion(s) plus an ablative margin), as assessed by CT, MRI, PET, US, and/or X-ray, at Visit 3 (between 7 days and less than 3 months post-ablation).
Target lesion recurrence (local recurrence) rate | 5 years post-ablation
  Target lesion recurrence (local recurrence) rate is evaluated at every visit after ablation of the target lesion(s), and overall evaluation at the 5-year follow-up, as assessed by CT, MRI, PET, US, and/or X-ray.

SECONDARY OUTCOMES:
Secondary efficacy rate | 5 years post-ablation
  Secondary efficacy rate, defined as the percentage of soft tissue lesions that have undergone successful repeat ablations (target or non-target) following identification of local soft tissue lesion progression, as assessed by CT, MRI, PET, US, and/or X-ray. A successful repeat ablation will be defined as ablation of the lesion according to the protocol and covered completely, with an adequate margin, as defined by the performing physician (i.e. the ablation zone completely overlaps or encompasses the lesion plus an ablative margin), as assessed by CT, MRI, PET, US, and/or X-ray, immediately following the procedure.
Regional recurrence rate at a separate location in the liver (outside the initial treatment site(s)) | 5 years post-ablation
  Regional recurrence rate at a separate location in the liver (outside the initial treatment site(s)), evaluated at every visit after ablation of the target lesion(s), and overall evaluation at the 5-year follow-up, as assessed by CT, MRI, PET, US, and/or X-ray.
Recurrence-free survival | 5 years post-ablation
  Recurrence-free survival, evaluated at every visit after ablation of the target lesion(s), and overall evaluation at the 5-year follow-up, as assessed by CT, MRI, PET, US, and/or X-ray.
Overall survival | 5 years post-ablation
  Overall survival, evaluated at every visit after ablation of the target lesion(s), and overall evaluation at the 5-year follow-up.
Economic impact of ablation as evaluated by complete procedure duration | Day of ablation (Day 0) through hospital discharge, estimated up to 1 week
Economic impact of ablation as evaluated by complete ablation duration | Day of ablation (Day 0) through hospital discharge, estimated up to 1 week
Economic impact of ablation as evaluated by number of ablations | Day of ablation (Day 0) through hospital discharge, estimated up to 1 week
Economic impact of ablation as evaluated by length of hospital stay | Day of ablation (Day 0) through hospital discharge, estimated up to 1 week
Economic impact of ablation as evaluated by number of probes used | Day of ablation (Day 0) through hospital discharge, estimated up to 1 week
Economic impact of ablation as evaluated by types of probes used | Day of ablation (Day 0) through hospital discharge, estimated up to 1 week
Incidence of reportable Adverse Events/Serious Adverse Events (AEs/SAEs) | 5 years post-ablation
  Incidence of adverse events (AEs) (SAEs) that are deemed at least unlikely related to the procedure or device and all serious adverse events (SAEs) from day of ablation through the end of the study.
Quality of Life Questionnaires (QLQ-C30 and QLQ-HCC18) | 9-12 months post-ablation
  European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 and liver-specific QLQ-HCC18 are questionnaires that will be completed at the Ablation Visit (pre-ablation), and each study visit afterwards, up to 9-12 months post-ablation.
  Note: These two questionnaires were chosen as tools to assess overall health status/quality of life in the patient population with soft-tissue liver lesions.
Numeric Pain Rating Scale | 7 days to 3 months post-ablation
  The Numeric Pain Rating Scale is a questionnaire where the patient reports their pain utilizing a 0-10 scale (where 0 is 'no pain' and 10 is 'maximum pain'). Patients will complete this questionnaire at the Ablation Visit (pre- and post-ablation), and at the first study visit after the ablation (7 days to 3 months post-ablation).

CONTACTS AND LOCATIONS:
Locations (28):
- United States (14):
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Olive View UCLA, Sylmar, California
  - Mayo Clinic, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin At Madison, Madison, Wisconsin
- China (2):
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
- France (2):
  - Hôpital Européen Georges-Pompidou, Paris
  - Tenon Hospital, Paris
- University Hospital Regensburg, Regensburg, Germany
- Netherlands (3):
  - VUMC Amsterdam, Amsterdam
  - University Medical Center Goningen, Groningen
  - Radboud UMC, Nijmegen
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Seoul National University Bundang Hospital (SNUBH), Seongnam-si, South Korea
- United Kingdom (3):
  - St. James's University Hospital, Leeds
  - The Royal Marsden Hospital, London
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu